CLINICAL TRIAL: NCT03276832
Title: Pilot Study to Test the Safety and Efficacy of the Combination of Imiquimod and Pembrolizumab for the Treatment of Metastatic Melanoma
Brief Title: Imiquimod and Pembrolizumab in Treating Patients With Stage IIIB-IV Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1578; NCI-2017-01591 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1578 (Other: Mayo Clinic in Florida); 16-002518 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Melanoma; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — Imiquimod; Biopsy; pembrolizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, imiquimod) (Experimental): Patients receive pembrolizumab IV on day 1 and apply imiquimod cutaneously on days 1-5 (Monday - Friday). Cycles repeat every 21 days for up to 2 years (approximately 35 courses) in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy at baseline, 6 weeks, and 12 weeks and CT, PET/CT, or MRI throughout the trial.
  Interventions: Drug: Imiquimod; Procedure: Biopsy; Biological: Pembrolizumab; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Imiquimod — Applied cutaneously
  Other Names: Aldara; R 837; S 26308; Zyclara
Procedure: Biopsy — Undergo biopsy
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; Nuclear Magnetic Resonance Imaging; NMRI; Structural MRI; sMRI

SUMMARY:
This pilot early phase I trial studies the side effects and how well imiquimod and pembrolizumab work in treating patients with stage IIIB-IV melanoma. Imiquimod may stimulate the immune system. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving imiquimod and pembrolizumab may work better at treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To gain preliminary data of the anti-tumor activity and safety profile of the combination of imiquimod and pembrolizumab in patients with unresectable cutaneous melanoma.

CORRELATIVE RESEARCH OBJECTIVES:

I. To compare and contrast (in a hypothesis generating manner) the biomarker profiles of patients who have a confirmed complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) criteria with patients who do not.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) on day 1 and apply imiquimod cutaneously on days 1-5 (Monday - Friday). Cycles repeat every 21 days for up to 2 years (approximately 35 courses) in the absence of disease progression or unacceptable toxicity. Patients undergo biopsy at baseline, 6 weeks, and 12 weeks and computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed up every 12 weeks for 1 year and then every 6 months for up to 3 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of stage IIIB, IIIC, IVM1a, IVM1b, or IVM1c that is not suitable for surgical resection
* Patients must not have received prior pembrolizumab or other anti-PD1/PDL1 therapies for their metastatic disease
* At least one cutaneous lesion that is amenable to treatment with topical imiquimod
* Measurable disease by RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 9.0 g/dL or >= 5.6 mmol/L without transfusion or (EPO) erythropoietin dependency (within 7 days of assessment)
* Serum total bilirubin =< 1.5 X upper limit of normal (ULN) or direct bilirubin =< (ULN) for subjects with total bilirubin levels > 1.5 ULN
* Aspartate transaminase (AST) =< 2.5 x ULN or =< 5 x ULN for subjects with liver metastases
* Albumin >= 2.5mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Creatinine =< 1.5 X upper limit of normal (ULN)

  * NOTE: measured or calculated (per institutional standard) creatinine clearance is acceptable >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Negative urine or serum pregnancy test done =< 72 hours prior to first treatment, for women of childbearing potential only

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Provide informed written consent
* Willing to return to enrolling institution for follow-up
* Willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion in appropriate low risk cutaneous lesions

  * NOTE: if the tissue biopsy is deemed to be of increased risk for the patient, the biopsy should not be performed and is optional
  * NOTE: newly-obtained is defined as a specimen obtained up to 42 days prior to registration where no anti-cancer therapy after the specimen was obtained and registration

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

    * NOTE: female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year; male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy; abstain from heterosexual activity is also acceptable method of contraception for males
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm or used an investigational device =< 4 weeks from registration
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Prior anti-cancer monoclonal antibody (mAb) =< 4 weeks prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks prior to registration
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy =< 2 weeks prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Known secondary malignancy that has progressed within the last 3 years or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Received a live vaccine =< 30 days prior to registration

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Duration of response | From registration to disease progression, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method.
Incidence of adverse events graded using Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years
  For each type of toxicity reported, the proportion of patients experiencing a severe level of that toxicity will be determined.
Overall survival | From registration to death due to any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method.
Progression free survival | From registration to documentation of first disease progression or death due to any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method.
Tumor response rate defined as percentage of patients whose objective disease status meets the criteria for Response Evaluation Criteria in Solid Tumors (RECIST) criteria for partial or complete response on two consecutive disease evaluations | Up to 2 years
  If there are no tumor responses documented among these 10 patients, then upper bound of a one-sided 95% confidence interval for the tumor response rate would be 25.9%.

SECONDARY OUTCOMES:
Biomarker changes during treatment | Baseline up to 12 weeks
  For each patient and each biomarker, a times-series plot of biomarker value will be constructed. These graphs will be visually examined for trends within and between the group of patients whose tumor responded to treatment and the group of patients whose tumor did not respond to treatment. Will include assessing total tumor RNA through RNA seq and PDL1 expression through the use of immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Ruqin Chen, MD, MB, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials